CLINICAL TRIAL: NCT01120275
Title: Phase II Study of RO4929097 (NSC-749225) in Advanced Melanoma
Brief Title: Gamma-Secretase/Notch Signalling Pathway Inhibitor RO4929097 in Treating Patients With Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02040; NCI-2011-02040 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0933; CDR0000671815; S0933 (Other: SWOG); S0933 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Acral Lentiginous Malignant Melanoma; Lentigo Maligna Malignant Melanoma; Nodular Malignant Melanoma; Recurrent Melanoma; Solar Radiation-related Skin Melanoma; Stage IV Melanoma; Superficial Spreading Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (gamma-secretase inhibitor RO4929097) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given PO
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well gamma-secretase/Notch signalling pathway inhibitor RO4929097 works in treating patients with stage IV melanoma. Gamma-secretase/Notch signalling pathway inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the six-month progression-free survival and one-year overall survival probability in Stage IV melanoma patients treated with RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097).

SECONDARY OBJECTIVES:

I. To investigate in a preliminary manner the relationship between Notch activation status and gene expression profile of tumor and clinical outcomes from patients in this study.

II. To study the effects of the investigational therapy on T cell function, which will provide a basis for subsequent trials combining Notch blockade with immunomodulatory therapy for advanced melanoma.

III. To assess the response rate (confirmed and unconfirmed complete and partial responses).

IV. To assess toxicity.

OUTLINE: This is a multicenter study.

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood collection at baseline and during study for analysis of T-cell function by flow cytometry and ELISA. Tumor tissue samples from biopsy or surgery are also analyzed for Notch activation by IHC and qRT-PCR.

After completion of study therapy, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed melanoma of cutaneous or unknown origin (ocular primary and mucosal primary excluded); patients must have Stage IV disease
* All patients must undergo a computed tomography (CT) or magnetic resonance imaging (MRI) of the brain within 42 days prior to registration that is negative for brain metastases; patients with a history of brain metastases are ineligible
* Patients must have measurable disease; all measurable lesions must be assessed (by physical examination, CT, or MRI scan) within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria In Solid Tumors [RECIST] 1.1); the CT from a combined positron emission tomography (PET)/CT must not be used to document measurable disease unless it is of diagnostic quality
* Sites must offer all patients participation in translational medicine studies and banking of paraffin embedded tissue and whole blood
* Patients must not have received any prior systemic therapy for Stage IV disease except for noncytotoxic biologic agents (e.g., vaccines, cytokines, cell therapies that do not require cytotoxic agents); patients may have received prior treatment with up to two prior biological therapies - no cytotoxics or kinase inhibitors - for advanced disease
* Patients may have had prior adjuvant immunotherapy with biological response modifiers (examples include but are not limited to interferon, vaccines, GM-CSF, and CTLA-4 blocking antibodies); prior adjuvant immunotherapy must have been completed at least 28 days prior to registration
* Adjuvant therapy containing cytotoxic agents is allowed if completed >= 180 days prior to registration
* Patients may have received prior radiation therapy; any side effects the patients had due to prior radiation therapy must have resolved to =< Grade 1 prior to registration; prior radiation therapy must have completed at least 28 days prior to registration
* Patients must have Zubrod performance status of 0-1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x IULN
* Serum creatinine =< IULN OR measured or calculated creatinine clearance >= 60 mL/min
* Patients must have the following serum electrolytes within the institutional ranges of normal: potassium, sodium, magnesium, phosphorous, chloride and calcium (corrected for serum albumin); these tests must be performed within 28 days prior to registration; patient must not require parenteral replacement therapy
* Patients must not have a history of allergic reaction attributed to compounds of similar chemical or biologic composition to RO4929097
* Patients must be able to swallow tablets
* Patients must not have malabsorption syndrome or other condition that would interfere with intestinal absorption of the agent
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin), are ineligible
* Patients must not be taking strong inducers or strong inhibitors of CYP3A4 at the time of registration
* Patients must not be known to be serologically positive for Hepatitis A, B, or C, or have a history of liver disease, other forms of hepatitis, or cirrhosis
* Patients must have an ECG within 28 days prior to registration. Patients must not have a QTcF > 450 msec (males) or QTcF > 470 msec (females)
* Patients must not have symptomatic congestive heart failure or unstable angina pectoris
* Patients with a history of torsades de pointes or any significant cardiac arrhythmia (except asymptomatic unifocal ventricular premature beats or supraventricular tachycardia easily controlled with oral medications) are excluded; any patient requiring or expected to require antiarrhythmics or other therapy known to prolong QTc is also excluded
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Women of childbearing potential must have a negative pregnancy test within 14 days prior to registration (the type of pregnancy test used is at the discretion of the registering institution); female patients of childbearing potential include the following:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Women must not be nursing due to possible harm to a nursing infant from the treatment regimen
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Margolin, Principal Investigator — SWOG Cancer Research Network
Locations (178):
- United States (178):
  - Providence Hospital, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Saint Edward Mercy Medical Center, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Tahoe Forest Cancer Center, Truckee, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Denver Veterans Administration Medical Center, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - University of Rochester, Rochester, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Adventist Medical Center, Portland, Oregon
  - SWOG, Portland, Oregon
  - AnMed Health Hospital, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Lee SM, Moon J, Redman BG, Chidiac T, Flaherty LE, Zha Y, Othus M, Ribas A, Sondak VK, Gajewski TF, Margolin KA. Phase 2 study of RO4929097, a gamma-secretase inhibitor, in metastatic melanoma: SWOG 0933. Cancer. 2015 Feb 1;121(3):432-440. doi: 10.1002/cncr.29055. Epub 2014 Sep 23. PMID 25250858

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Gamma-secretase Inhibitor RO4929097)
Started | 36
Eligible and Treated | 32
Completed | 0
Not Completed | 36
Not completed — Adverse Event | 3
Not completed — Progression | 27
Not completed — Ineligible | 3
Not completed — Withdrawal by Subject | 1
Not completed — Refusal | 1
Not completed — Not specific | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who had received the protocol treatments were included in the baseline analysis.
Arm/Group | Treatment (Gamma-secretase Inhibitor RO4929097)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 60.9 [32.8 to 85.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Performance Status [Number; unit: participants] — Patients were graded according to the Zubrod Performance Status Scale. Performance Status is 0 if patient is fully active, able to carry on all pre-disease performance without restriction. Performance Status is 1 if patient is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0 | 24
    1 | 8
Primary Type [Number; unit: participants]
  Cutaneous | 22
  Unknown primary | 10
Site(s) of Metastases [Number; unit: participants] — Distant metastatic involvement is defined as the presence of one or more metastases beyond the regional lymph node drainage.
  participants
    Bone | 8
    Liver | 12
    Lymph node, skin, soft tissue | 17
    Lung | 17
    Other non-visceral | 1
    Other visceral | 9
Elevated Lactate Dehydrogenase (LDH) [Number; unit: participants]
  No | 19
  Yes | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause.
Time Frame: Disease assessments were performed every 6 weeks, up to 3 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Gamma-secretase Inhibitor RO4929097)
Number analyzed (Participants) | 32
Months | 1.5 [1.3 to 2.6]
Statistical Analysis 1: Comparison: Treatment (Gamma-secretase Inhibitor RO4929097); 6-month progression free survival (PFS) was estimated using the method of Kaplan-Meier and confidence intervals were calculated using the log-log transformation; Test type: Superiority or Other; 6-month PFS = 0.09, 95% CI 2-sided [0.02 to 0.22]

2. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Weekly, up to 3 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Gamma-secretase Inhibitor RO4929097)
Number analyzed (Participants) | 32
Months | 13 [8 to 20]
Statistical Analysis 1: Comparison: Treatment (Gamma-secretase Inhibitor RO4929097); 1-year overall survival (OS) was estimated using the method of Kaplan-Meier and confidence intervals were calculated using the log-log transformation; Test type: Superiority or Other; 1-year OS = 0.5, 95% CI 2-sided [0.32 to 0.66]

3. Secondary Outcome: Percentage of Participants With Confirmed and Unconfirmed Complete or Partial Response
Description: Complete disappearance of all measurable and non-measurable disease, or greater than or equal to 30% decrease under baseline of the sum of the longest diameters of all target measurable lesions.
Time Frame: Disease assessments for response were performed every 6 weeks, up to 3 years
Measure: Number (95% Confidence Interval); unit: portation of participants
Arm/Group | Treatment (Gamma-secretase Inhibitor RO4929097)
Number analyzed (Participants) | 32
portation of participants | 0.03 [0 to 0.16]

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment was evaluated at least every 3 weeks at the beginning of each cycle, up to 3 years
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- RO4929097: Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | RO4929097
Number analyzed (Participants) | 32
Participants
  Abdominal pain | 1
  Alanine aminotransferase increased | 1
  Anemia | 1
  Electrocardiogram QT corrected interval prolonged | 1
  Fatigue | 1
  Hypophosphatemia | 2
  Lymphocyte count decreased | 1
  Nausea | 1
  Pain in extremity | 1
  Small intestinal obstruction | 1
  Stroke | 1

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated at least every 3 weeks at the beginning of each cycle, up to 3 years.
Description: Per protocol, Grade 4 myelosuppression does not require expedited reporting via the NCI's Adverse Event Expedited Reporting System (AdEERS). The protocol does not specify that all AEs Gr 3 and higher require expedited reporting.
Groups:
- RO4929097: Patients receive gamma-secretase/Notch signaling pathway inhibitor RO4929097 PO on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | RO4929097
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO4929097 (N=32)
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO4929097 (N=32)
Anemia (Blood and lymphatic system disorders) | 7
Sinus bradycardia (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 16
Pain (General disorders) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 5
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less